CLINICAL TRIAL: NCT06406751
Title: Microbiome Effects of Extended Use of MI Paste in Elderly Removable Denture Wearers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Robert Bowers, Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202401429
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Dental Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MI Paste Application for 14 days (Experimental): Subjects will apply 1 cubic centimeter of MI Paste for 14 days.
  Interventions: Device: MI Paste

INTERVENTIONS:
Device: MI Paste — Sterile swabs will be used to collect plaque from under the subject's upper denture (when the denture is removed) and the subject's mouth tissues. This will be used for genomic DNA, bacteria analysis, and fungus analysis. Subjects will also apply 1 cubic centimeter of MI Paste to the fitting surface on a daily basis for 14 days. Afterward, subjects will return to the clinic for another sterile swab to be collected.

SUMMARY:
The purpose of this study is to determine if MI Paste affects the bacteria and fungus present within the mouth, as well as to determine if MI Paste increases denture comfort and retention. MI Paste is a water-based topical dental product that is available without a prescription. It is generally used to treat dental/tooth hypersensitivity (sensitive teeth) in patients and/or to help re-mineralize the tooth enamel in patients. Within this study, there is an off-label use for research subjects to apply above the upper denture.

DETAILED DESCRIPTION:
Potentially-eligible subjects will be invited to the research study that involves consenting and 4 in-person visits (Screening Visit, Visit 1, Visit 2, Visit 3) where the following will be performed at each visit: (i) upper denture/mouth tissues swab sample collected, (ii) survey questions being administered, and (iii) brief oral dental exam (clinical assessment). Furthermore, at Visit 2, subjects will be provided and instructed on how to use MI Paste under their removable upper denture for 14 days and instructed to monitor symptoms of comfort, retention, and dry mouth (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 65 years of age,
* Capacity to independently provide consent,
* Having an adequately fitting removable complete maxillary (upper jaw) denture (no consideration relative to the presence or type of mandibular prosthesis (lower jaw partial or full denture).

Exclusion Criteria:

* ill-fitting complete denture(s),
* presence of pathology indicated for immediate treatment (epulis fissuratum (excess folds of firm tissue form inside the mouth, as a result of rubbing on the edge of dentures that do not fit well), large denture sores),
* currently or previously taking any form of antibiotics or antifungals (oral, intravenous, mouthwashes) over the previous two months that may impact microbial assessments.
* a history of food-based allergies: casein, lactose, or food/cosmetic ingredient preservatives. These exclusions have been made out of an abundance of caution to avoid any potential adverse reaction to MI Paste which contains casein phosphopeptide--amorphous calcium phosphate (CPP-ACP), and several common preservative ingredients in oral care products that may induce sensitivities/allergic reaction in a small portion of the population.
* milk allergy

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in the oral microbiome composition over time | Multiple time points (baseline, two weeks, and four weeks)
  16S genomic profiling will be done in all recruited subjects via oral swab from under the denture and mouth tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bowers, DDS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Dentistry, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No